CLINICAL TRIAL: NCT06384456
Title: The Effect of Topical TRanexamic Acid Vs. Placebo on Acute Postoperative Pain Following Distal Radius Fracture Fixation: a Randomized Controlled Trial - the TRADR Study
Brief Title: Topical TRanexamic Acid Vs. Placebo on Acute Postoperative Pain Following DRF Fixation
Acronym: TRADR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ryan Paul, Dr., University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-5708
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fractures
Keywords: Distal Radius Fractures; acute pain; Topical tranexamic acid; Open Reduction and Internal FIxation; Placebo; Randomized Control Trial
MeSH Terms: conditions — Wrist Fractures; Acute Pain | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical TRanexamic Acid (Experimental): 10mL of 100mg/mL TXA in addition to the standard care
  Interventions: Drug: Topical TRanexamic Acid
- Placebo (Placebo Comparator): 10mL of 100mg/mL normal saline in addition to the standard care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical TRanexamic Acid — 10mL of 100mg/mL TXA will be administered into the surgical wound prior closure.
  Arms: Topical TRanexamic Acid
Drug: Placebo — 10mL of 100mg/mL normal saline will be administered into the surgical wound prior closure.
  Arms: Placebo

SUMMARY:
The goal of this study is to find out whether the use of topical tranexamic acid (TXA) into the surgical wound will result in less post-operative pain, less pain killer use, and better post-operative use of the wrist in people undergoing surgery for a wrist fracture compared to not using topical TXA (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open reduction internal fixation (Volar approach) for operative management of a distal radius fracture;
* Aged 18 or older;
* Provision of informed consent;
* Cognitive ability and English-language skills required to complete outcome measures.

Exclusion Criteria:

* Revision surgery or any additional operative management of ipsilateral wrist injury
* Distal radius fracture treated with a dorsal approach
* Known history of lymphedema or lymph node dissection in the operative extremity
* Known chronic pain conditions, fibromyalgia, or polymyalgia rheumatic
* Current user of opioids and/or on chronic opioids use
* Known allergic reaction to TXA
* Anticoagulant use not stopped in time for surgery as per thrombosis Canada guidelines (i.e. warfarin, acetylsalicylic acid, direct oral anticoagulants, etc.)
* Previous thrombotic stroke or thromboembolic disorders (i.e. known previous DVT, PE, or clotting disorders)
* Current pregnancy or breastfeeding
* Previous neurologic injury causing paralysis of affected shoulder/arm
* Severe cardio-respiratory disease (i.e. ASA Grade IV or higher).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
acute post-op pain | 24 hours to 72 hours postoperatively
  It will be assessed with VAS 0 to 10cm, with higher score indicating worse pain.

SECONDARY OUTCOMES:
opioid use | 1, 2, and 6-week post-surgery
  Opioid use will be recorded on patients' medication diary
persistent pain | 1, 2, and 6-week post-surgery
  It will be assessed with VAS 0 to 10cm, with higher score indicating worse pain.
unscheduled hand-related procedures | 1, 2, and 6-week post-surgery
  clinic/emergency unit visits or any issue or events related to the condition that might lead participant to visit the emergency room, be seen by a doctor, or undergo any intervention more frequently than the usual visits
Patient reported function | 1, 2, and 6-week post-surgery
  will be assessed using the disabilities of the arm, shoulder and hand questionnaire (DASH) score 0 to 100, with higher score indicating more disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lameire DL, Noori A, Abbas A, Persitz J, Baltzer H, Collett E, Veillette C, Chan A, Paul R. The effect of topical TRanexamic Acid versus placebo on acute postoperative pain following Distal Radius fracture fixation: protocol for a randomised controlled trial at a quaternary care hand surgery centre - The TRADR study. BMJ Open. 2025 May 21;15(5):e095684. doi: 10.1136/bmjopen-2024-095684. PMID 40398932